CLINICAL TRIAL: NCT04314557
Title: Renal Arterial Denervation in Sympathetic Dysautonomia: RANSOM REGISTRY
Brief Title: Renal Arterial Denervation in Sympathetic Dysautonomia
Acronym: RANSOM
Status: Completed | Type: Observational
Sponsor: St Carlos Hospital, Madrid, Spain (Other)
Responsible Party: Principal Investigator, IVAN J NUÑEZ GIL, Principal Investigator. Attending Physician. MD, PhD, FESC, St Carlos Hospital, Madrid, Spain
Other Study IDs: 18/532-O_P
Record Dates: First submitted 2019-12-16; First posted 2020-03-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Renal Denervation; Increased Variability; Blood Pressure Disorders; Blood Pressure Variability; Sympathetic Dysautonomia
Keywords: Sympathetic dysautonomia; Blood Pressure Variability; Hypertension; Renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Renal denervation — Spyral device. Bilateral renal denervation.

SUMMARY:
The RANSOM registry is considered as a collection of data with the ultimate purpose of gathering information about the effect of renal denervation in patients of the investigator's center and evaluating the results within the usual clinical practice.

The general objective of the study is to evaluate the clinical results (blood pressure, quality of life and levels of catecholamines) as well as safety of renal sympathetic denervation in hypertensive patients, at least in treatment with an antihypertensive drug and with increased variability, considering as such a standard deviation> 10 mmHg for systolic BP and> 5 for diastolic BP of its blood pressure levels, measured by ABPM.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in a prospective manner must sign an informed written consent and meet ALL of the following criteria that are typical of the procedure according to the protocol of our center:
* Be considered adequate and eligible by the group of doctors responsible for the patient and by the multidisciplinary team of the study. Over 18 years, not pregnant.
* Poorly controlled arterial hypertension, under treatment with at least one antihypertensive drug.
* In addition, poorly controlled hypertension + increased variability, considering as such a standard deviation> 10 mmHg for systolic BP and> 5 for the diastolic BP of patient´s blood pressure levels, measured by ABPM.
* Renal arteries anatomy suitable for the procedure, considered by CT, MRI, ultrasound or angiography.
* Some criteria of dysautonomia, following the consensus of the American Autonomous Society (AAS) and the European Federation of Autonomous Societies (EFAS) of 2018.

or supine HTN. Defined as sBP ≥ 140 mmHg and / or dBP ≥ 90 mmHg, measured at least after 5 minutes of supine rest. Moderate forms (160-179 mmHg or dBP of 100-109 mmHg) or severe will preferably be included. (sBP≥ 180 mmHg and / or dBP ≥ 110 mmHg). Mild forms will be considered in conjunction with symptoms or other findings (ABPM) or nighttime HTN. Considered as such one that does not fall more than 10% compared to the daytime BP or even rises (riser). They will be considered in conjunction with symptoms or other findings (eg ABMP).

* If the foregoing is not fulfilled, marked orthostatism (> 30 mmHG in sBP and / or> 10mmHG in dBP).
* Life expectancy exceeding one year (not presenting terminal illness or any health condition for which a survival of less than one year is estimated).

Exclusion Criteria:

* eGFR <30 mL / min / 1.73m2.
* Monoxidin treatment.
* Impossibility of informed consent by the patient or legal representative.
* Impossibility for follow-up at least 1 year.
* Do not fulfill inclusion criteria, assessed by the multidisciplinary team.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the descent of Systolic BP in orthostatism | 12 months
  BP Variability decrease, any (yes/no).

SECONDARY OUTCOMES:
Change in the descent of Systolic BP in orthostatism. | 12 months
  BP Variability decrease < 25 percent (yes/no)
Measurement of quality of life and subjective perception of well-being. | 12 months
  Short form 12, questionaire (0-100, the higher the better).
Evolution of blood pressure control, average levels and variability | 12 months
  AMPA measure mean PA levels (numeric)
Safety end points | 12 months
  MACE (death,bleeding, renal failure-yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Catala-Lopez F, Sanfelix-Gimeno G, Garcia-Torres C, Ridao M, Peiro S. Control of arterial hypertension in Spain: a systematic review and meta-analysis of 76 epidemiological studies on 341 632 participants. J Hypertens. 2012 Jan;30(1):168-76. doi: 10.1097/HJH.0b013e32834d30ec. PMID 22025240
- [Background] Kotseva K, De Bacquer D, De Backer G, Ryden L, Jennings C, Gyberg V, Abreu A, Aguiar C, Conde AC, Davletov K, Dilic M, Dolzhenko M, Gaita D, Georgiev B, Gotcheva N, Lalic N, Laucevicius A, Lovic D, Mancas S, Milicic D, Oganov R, Pajak A, Pogosova N, Reiner Z, Vulic D, Wood D, On Behalf Of The Euroaspire Investigators. Lifestyle and risk factor management in people at high risk of cardiovascular disease. A report from the European Society of Cardiology European Action on Secondary and Primary Prevention by Intervention to Reduce Events (EUROASPIRE) IV cross-sectional survey in 14 European regions. Eur J Prev Cardiol. 2016 Dec;23(18):2007-2018. doi: 10.1177/2047487316667784. Epub 2016 Sep 27. PMID 27638542
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Hering D, Grassi G. Effects of renal denervation on short-term blood pressure variability: lack of meta-analytic evidence. J Hypertens. 2017 Sep;35(9):1780-1781. doi: 10.1097/HJH.0000000000001397. No abstract available. PMID 28767486
- [Background] Fanciulli A, Jordan J, Biaggioni I, Calandra-Buonaura G, Cheshire WP, Cortelli P, Eschlboeck S, Grassi G, Hilz MJ, Kaufmann H, Lahrmann H, Mancia G, Mayer G, Norcliffe-Kaufmann L, Pavy-Le Traon A, Raj SR, Robertson D, Rocha I, Struhal W, Thijs R, Tsioufis KP, van Dijk JG, Wenning GK. Consensus statement on the definition of neurogenic supine hypertension in cardiovascular autonomic failure by the American Autonomic Society (AAS) and the European Federation of Autonomic Societies (EFAS) : Endorsed by the European Academy of Neurology (EAN) and the European Society of Hypertension (ESH). Clin Auton Res. 2018 Aug;28(4):355-362. doi: 10.1007/s10286-018-0529-8. Epub 2018 May 15. PMID 29766366
- [Background] Núñez-Gil IJ. Protocolo Asistencial de denervación renal percutánea mediante radiofrecuencia. Hospital Clínico San Carlos 2016.
- [Background] Nunez-Gil IJ, Garcia-Donaire JA, Vedia O, Abad-Cardiel M, Martell-Claros N, Fernandez-Ortiz A. [Initial experience with a multi-electrode catheter in renal denervation. A technique that has come back to stay?]. Hipertens Riesgo Vasc. 2019 Jul-Sep;36(3):166-168. doi: 10.1016/j.hipert.2019.04.002. Epub 2019 May 31. No abstract available. Spanish. PMID 31160234
- [Background] Travieso-Gonzalez A, Nunez-Gil IJ, Riha H, Donaire JAG, Ramakrishna H. Management of Arterial Hypertension: 2018 ACC/AHA Versus ESC Guidelines and Perioperative Implications. J Cardiothorac Vasc Anesth. 2019 Dec;33(12):3496-3503. doi: 10.1053/j.jvca.2019.03.068. Epub 2019 Apr 3. PMID 31078374
- See also: Spyral device description/label — https://manuals.medtronic.com/manuals/main/en_ES/manual/index